CLINICAL TRIAL: NCT06632210
Title: Psychological Effects of Helicopter Pylori Associated Gastritis in Patients Attending Assiut University Hospitals
Brief Title: Psychological Effects of H Pylori Associated Gastritis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ashraf khalifa Darweesh Desokey, Principal investigator, Assiut University
Other Study IDs: H pylori associated gastritis
Record Dates: First submitted 2024-09-30; First posted 2024-10-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: H Pylori

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goals of this study

1. Explore association between psychological factors and Hpylori associated gastritis.
2. Assess prevalence and severity of psychology symptoms among patients with H pylori associated gastritis and their effects on their life.
3. Examine relation between demographic and clinical variables .
4. Effect of eradication of H pylori on psychological status of patients.

DETAILED DESCRIPTION:
One of the most prevalant chronic bacterial illness affecting people is it H.plyori infection. it affects at least 50% of people worldwide . it is a human gastrointestinal infection which is believed to be blammed for a number of gastric illness from chronic gastritis up to gastric cancer.

numerous literature data suggest there is strong relation of anxiety disorders, stress or depression to somatic symptoms and this relation can undergo potentialization in case of appearance of pathogenic factors like helicobacter pylori infection , this relation can confirmed with many scientific reports , with the common use of antidepressants and anxiety relieving drugs in duodenal ulcer disease therapy.

The close relationship of gastrointestinal function with brain function and the mental status is known as (gut brain axis).

it has been reported that emotional factors induce changes in gastric physiology that physiological stress induces personality dependant gastric acid secretion changes and avariety of alterations in gastric motility.

. the effect of numerous stress factors which injury mucosa of stomach and modify immunity of the patient so that the patient become more sensitive to be infected with H. Pylori and infection become more aggressive and lead to manifestation of gastritis , duodenitis and gastric ulcer disease.

mental stress is considered a major pathogenic factor for peptic ulcers and it is associated with increasing prevalence of gastric ulcersin patients is with or without H.pyloriinfection.

another study revealed that depression is associated with food related symptoms as nausea and vomiting ,similarly it was showing that gastric information lead to an anxiety and depression like behaviors via neuroendocrine pathways in female not male.

so the investigetors conducted this observational study to determine the most common physiological effect is of H.pylori associated gastritis in patients attending Assiut university hospitals and How to deal with it to improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. all patients with H.Pylori associated gastritis that diagnosed by endoscopy.
2. patients diagnosed by detection of H.Pylori Ag in stool

Exclusion Criteria:

1. patients did not take antibiotics within last 2 weeks
2. patients did not take PPI within last 1 month
3. patients not with acute massive GITbleeding.
4. patients without eradication of H.Pylor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * all patients with H.Pylori associated gastritis that diagnosed by endoscopy.
  * patients diagnosed by detection of H.Pylori Ag in stool
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2026-03-22 (Estimated); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
The aim of this observational study is to Explore correlation between psychological factors and H.Pylori associated gastritis . | 2024
  The aim of this observational study is to Explore correlation between psychological factors and H.Pylori associated gastritis .

CONTACTS AND LOCATIONS:
Overall Officials: Nabila fayeg Amen, Professor, Study Director — Assiut University; Mohammed Abozaid Ali, Doctor, Study Director — Assiut University